CLINICAL TRIAL: NCT00430170
Title: Does Caffeine Reduce Dipyridamole-Induced Protection Against Ischemia-Reperfusion Injury?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: G Rongen, dept Pharmacology Toxicology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dipy001
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Cardiovascular Disease; Ischemia-Reperfusion Injury
Keywords: ischemia-reperfusion injury; adenosine; dipyridamole; caffeine
MeSH Terms: conditions — Cardiovascular Diseases; Reperfusion Injury | interventions — Dipyridamole; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): dipyridamol during 7 days and before ischemic exercise caffeine 4mg/kg
  Interventions: Drug: Dipyridamole; Drug: caffeine
- 2 (Placebo Comparator): dipyridamol during 7 days and before ischemic exercise placebo
  Interventions: Drug: Dipyridamole

INTERVENTIONS:
Drug: Dipyridamole — Dipyridamole 2x200mg 7day per os
  Other Names: persatin
Drug: caffeine — caffeine 4mg/kg iv
  Arms: 1

SUMMARY:
The purpose of this project is to explore the interaction between caffeine and dipyridamole on ischemia-reperfusion injury in the forearm.

DETAILED DESCRIPTION:
Dipyridamole has been proven to reduce targeting of Annexin A5 in responses to ischemic exercise, indicating protection against ischemia-reperfusion injury in humans (pharmacological preconditioning). Dipyridamole increases the endogenous adenosine level by inhibition of the nucleoside transporter (ENT-1). Activation of the adenosine receptor protects against ischemia-reperfusion injury. We hypothesize that endogenous adenosine mediates the protective effect of dipyridamole against ischemia-reperfusion injury. Therefore the adenosine receptor antagonist caffeine will reduce the benefit of dipyridamole on forearm ischemia-reperfusion injury.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 18-50yr.

Exclusion Criteria:

* cardiovascular disease
* hypertension (systole > 140 mmHg, diastole > 90 mmHg)
* hypercholesterolemia (random total cholesterol > 6.5 mmol/l)
* diabetes mellitus (fasting glucose > 7.0 mmol/L or random glucose > 11.0 mmol/L)
* asthma (recurrent episodes of dyspnea and wheezing, or usage of prescribed inhalation medication: i.e. corticosteroids or B2-agonists)
* participation in any clinical trial during the last 60 days prior to this study.
* administration of two doses of Annexin A5 (0,1mg; 450MBq) during the last 5 years prior to this study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Percentage difference in Annexin A5 targetting between experimental and control thenar muscle at 60 and 240 minutes after reperfusion | 60 and 240 minutes after ischemic exercise

SECONDARY OUTCOMES:
Plasma dipyridamole concentration | at the morning of day 7 of treatment with dipyridamole/placebo
ENT transport activity (before and after treatment with dipyridamole 200mg, twice daily, for seven days) | before start of treatment (dipyridamol/placebo) and in the morning of day 7 of treatment (placebo/dipyridamol)
Workload (duration of exercise and developed force) | during 10 minutes of ischemic exercise

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Riksen NP, Oyen WJ, Ramakers BP, Van den Broek PH, Engbersen R, Boerman OC, Smits P, Rongen GA. Oral therapy with dipyridamole limits ischemia-reperfusion injury in humans. Clin Pharmacol Ther. 2005 Jul;78(1):52-9. doi: 10.1016/j.clpt.2005.03.003. PMID 16003293
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546